CLINICAL TRIAL: NCT04567992
Title: Efficacy of Ultrasound Guided Superficial Cervical Plexus Block for Tracheal Reconstruction Surgery on Quality of Recovery: a Randomized Control Study
Brief Title: Efficacy of Ultrasound Guided Superficial Cervical Plexus Block for Tracheal Reconstruction Surgery:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ayman Abougabal, lecturer of anaesthesia, SICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-106-2020
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2020-10

CONDITIONS: Efficiency of Using Ultrasound-guided SCB for Providing Intra and Postoperative Analgesiatracheal Reconstruction Surgery
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCPB (Experimental)
  Interventions: Procedure: superficial cervical plexus block
- Control (Placebo Comparator)
  Interventions: Procedure: superficial cervical plexus block

INTERVENTIONS:
Procedure: superficial cervical plexus block — ultrasound guided injection of local anaesthesia in the superficial cervical plexus
  Other Names: Drug:; Bupivicaine

SUMMARY:
The essential goal for tracheal reconstruction is is the ability of the anaesthesiologist and surgeon to maintain control of the airway at all times. In the postoperative period the patient should maintain a flexed neck position to avoid any traction on the tracheal anastomosis. Thus, pain control is essential postoperatively so that patients will be awake and cooperative to maintain this position. [1].

Superficial cervical plexus block can be used in a variety of surgical procedures , including superficial surgery on the neck and shoulders and thyroid surgery as it results in anesthesia of the skin of the anterolateral neck and the ante-auricular and retro-auricular areas, as well as the skin overlying and immediately inferior to the clavicle on the chest wall Figures 1 and 6)[2].

Thus it can be used as an adjuvant to general anaesthesia to provide analgesia for patients undergoing tracheal resection and anastomosis to keep the patients awake and cooperative at the conclusion of the procedure.

The goal of the ultrasound (US)-guided technique of SCB is to deposit local anesthetic within the vicinity of the sensory branches of the nerve roots C2, C3, and C4 which combine to form the four terminal branches (the lesser occipital, greater auricular, transverse cervical, and supraclavicular nerves) and emerge from behind the posterior border of the SCM. Advantages over the landmark-based technique include the ability to visualize the spread of local anesthetic in the correct plane, which therefore increases the success rate, and to avoid a needle insertion that is too deep and the inadvertent puncture of neighboring structures[3].

Aim of the work To assess the efficiency of using ultrasound-guided SCB for providing intra and postoperative analgesia for patients undergoing tracheal resection and anastomosis under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

• ASA physical status I, II, and III adult patients undergoing elective tracheal resection and anastomosis under general anaesthesia were included.

Exclusion Criteria:

* Coagulation disorders
* Pregnancy.
* Age less than 18 years.
* Patient refusal.
* Emergency re-operation within

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
quality of recovery using quality of recovery 40 qusetionnaire | first 24 hour
  total score of Qor-40 (total score of 200) with highest indicates better outcome

SECONDARY OUTCOMES:
post operative morphine consumption | 24 hour
  post operative morphine consumption
visual analogue scale post-operative | first 24 hour
  visual analogue scale post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No